CLINICAL TRIAL: NCT02672982
Title: Follow Up of Severely Malnourished Children (FUSAM): Effectiveness of a Combined Nutrition Psychosocial Intervention on Health and Development.
Brief Title: Follow Up of Severely Malnourished Children (FUSAM)
Acronym: FUSAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Action Contre la Faim (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACFInternational
Record Dates: First submitted 2015-01-13; First posted 2016-02-03 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Severe Acute Malnutrition
Keywords: Severe acute malnutrition; Psychosocial intervention; Child; Stimulation; CMAM; Nepal
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- new combined NUTPSY treatment (Experimental): 2-month combined nutrition and psychosocial intervention
  Interventions: Other: NUTPSY treatment
- standard NUT treatment (Active Comparator): 2-month of standard nutritional treatment only
  Interventions: Other: NUT treatment

INTERVENTIONS:
Other: NUTPSY treatment — The psychosocial component of the new combined treatment involves seven weekly counselling sessions with mothers focused on feeding, emotional attachment, stages of child development, stimulation, emotional responsiveness and interaction, and on concerns/strategies of child care and parenting.
  Arms: new combined NUTPSY treatment
Other: NUT treatment — Only the standard nutritional treatment in the form of Ready-to-use Therapeutic Food (RUTF) is administered.
  Arms: standard NUT treatment

SUMMARY:
The overall objective of the research is to assess the long-term and cost-effectiveness of a combined nutrition psychosocial intervention to a stand-alone nutritional treatment of children with Severe Acute Malnutrition (SAM) aged 6 to 24 months in the Saptari District of Nepal.

DETAILED DESCRIPTION:
In Nepal, the majority of SAM children are treated with therapeutic food in community/home-based care, and little is known about the long-term sustainability of the nutritional and health benefits of treatment after rehabilitation. The two treatments will be compared in terms of costs of treatment and convened health benefits (child nutritional status and development, cured rate and relapse, maternal mental health, and family care practices) at both short and long-term periods after admission. The proposed complementary psychosocial intervention focuses directly on the key underlying determinants of acute malnutrition within children's early years, such as child care practices and stimulation, parent-child relationships and maternal mental health. It includes the mother/caregiver as patient of psychosocial support, but also empowers her as the key ally in the treatment of the undernourished child. Adding a brief psychosocial component to the standard medico-nutritional treatment is expected to pay off in terms of sustainable recovery, health, and development outcomes of children.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-23 months
* 2 sexes
* Diagnosis: uncomplicated severe acute malnutrition requiring follow-up outpatient therapeutic feeding unit (OTPs), supported by Action Contre la Faim in Saptari district
* Weight-for-height (WH) <-3 Standard Deviation compared to the WHO reference and/or MUAC <115 mm
* And / or nutritional oedema moderate (+ or + +)
* And successful test of appetite
* And no medical complications
* New cases
* Presence of mother / father or legal guardian aged > 18 years.
* Understanding of the consent and information letter
* Follow-up possible

Exclusion Criteria:

* Age <6 months or> 24 months
* Moderate Acute Malnutrition
* Severe Acute Malnutrition complicated
* Weight for height <-3 Standard Deviation compared to the WHO reference and / or MUAC <115mm but failure to test appetite OR medical complications OR severe oedema + + + OR kwashiorkor, marasmus (malnutrition with the same criteria, with oedema mild or severe).
* Relapse or if already registered in the past two months;
* Any child with developmental anomalies, known chronic illnesses like epilepsy, twins and multiple births, parents not consenting,

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 427 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Child motor, cognitive, emotional and social development assessed with Ages and Stages Questionnaire | up to 11 months after inclusion
  The Ages and Stages Questionnaire (Squires et al, 1999), is a low-cost, easily administered, parent-report screening test of development in communication, motor, problem-solving and personal-social domains. The questionnaire has been adapted and used in low- and middle-income countries in Africa, Asia and Latin America, where it has demonstrated sensitivity to child nutritional status and psychosocial stimulation. While it is not a diagnostic test, it offers an opportunity to systematically obtain information about children's development with an instrument that does not require extensive training

SECONDARY OUTCOMES:
Child Care Practices | Up to 11 months after inclusion
  The quality of care practices is measured by assessing the level of knowledge and the practices. It comprises sub-thematics: care for women, pregnancy and delivery, care for the newborn, breastfeeding and feeding, access to resources for care, as well as child development and psychosocial care. The Child Care Knowledge & Practices Questionnaire has been developped by Action Contre la Faim.
Mother-child interaction | Up to 11 months after inclusion
  Action Contre la Faim's Mother-Child Interaction Grid will be used for assessing the quality of mother-child interactions and interpersonal sensitivity and responsiveness.
Child stimulation | Up to 11 months after inclusion
  Family Care Indicators (FCI) (Frongillo et al, 2003) is used to assess the quality of child stimulation
Maternal perinatal mental health | Up to 11 months after inclusion
  The Edinburgh Post-natal Depression Scale (Cox et al, 1987) is a valuable and efficient way of identifying mothers at risk for "perinatal" depression.
Perceived Social Support | Up to 11 months after inclusion
  The Multidimensional Scale of Perceived Social Support (Zimet et al, 1988) measures perceived support from 3 sources: family, friends and significant others.
Maternal self-esteem | Up to 11 months after inclusion
  The Rosenberg self-esteem scale (Rosenberg, 1965) assesses maternal self-esteem.
Maternal mental health | Up to 11 months after inclusion
  The WHO Self Reporting Questionnaire (SRQ-20) (WHO, 1994) assesses the frequency of depressive symptoms, anxiety, and psychosomatic complaints in the past month. The measure has been shown to be an accurate predictor of common mental disorder and has been successfully used in several studies in developing countries.
Child growth (height) | Up to 11 months after inclusion
  Child growth measures change in height
Child nutritional status defined by Mid-Upper Arm Circumference (MUAC) | Up to 11 months after inclusion
  Comparison of the mean MUAC adjusted to age, sex and height
Child nutritional status defined by Weight-For-Height Z-score | Up to 11 months after inclusion
  Comparison of the mean Weight-For-Height Z-score
Child nutritional status defined by height-for-Age Z score | Up to 11 months after inclusion
  Comparison of the mean height-for-Age Z score
Child health status (morbidity rate) | Up to 11 months after inclusion
  Follow-up of morbidity rate
Child death (mortality rate) | Up to 11 months after inclusion
  Follow-up of mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Bizouerne, PhD, Principal Investigator — Action Contre la Faim
Locations (1):
- ACF, Nepal, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Media link from the first communication event of the FUSAM project in Nepal and steering committee meeting — http://www.spotlightnepal.com/News/Article/UNDER-NUTRITION-ACF-Follow-Up-Works
- See also: Oral presentation at the ACF International conference in Nepal, June 2017 — https://acfinternationalconference2017.wordpress.com/oral-presentations/